CLINICAL TRIAL: NCT00713375
Title: Multiscale Entropy and Time-Frequency Analysis of Electrocardiogram and Blood Pressure in Patients With Spontaneous Intracranial Hemorrhage
Brief Title: Time Frequency Analysis of Electrocardiogram and Blood Pressure in Intracranial Hemorrhage Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Kuo-Chuan Wang, MD, National Taiwan University Hospital
Other Study IDs: 200803013R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Subarachnoid Hemorrhage; Intracranial Hemorrhages; Cerebral Hemorrhage
Keywords: Autonomic Nervous System; Subarachnoid Hemorrhage; Intracranial Hemorrhages; Cerebral Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Hemorrhages; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood. Cerebral spinal fluids
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Dysregulation of autonomic nervous system is evident in patients with spontaneous intracranial hemorrhage. In this study, we utilize a non-invasive method (heart rate and blood pressure variability analysis to analyze the autonomic activities in this group of neurosurgical patients. Our aim is to determine the utility of this modality in risk stratification and outcome prediction in these patients.

DETAILED DESCRIPTION:
Spontaneous intracranial hemorrhage is an absolute emergency in the field of neurosurgery, and it is also a devastating event that commonly results in major neurological disabilities or mortalities. Since disease severities and clinical courses vary in each patient, pathophysiological studies and prognostic factors are always worth research. From previous studies, we know that dysregulation of autonomic system plays an important role in intracranial hemorrhage. Hemorrhage itself is associated with sympathoexcitation, and patients who develop rebleeding or infarction complications are found to have an even higher degree of sympathetic storm. Therefore, the degree of autonomic activities seems to be a useful predictor.

Traditionally, sympathetic activities are measured by plasma catecholamine, while parasympathetic activities are hard to measure. In recent decades, the application of engineering in biological fields makes a great breakthrough. Waveform analysis of biological signals, such as electrocardiograms and arterial blood pressure, can indirectly determine autonomic activities. The variabilities of heart rate and blood pressure are subjected to frequency analysis. This generates several dominant frequency bands. High frequency bands (0.15-0.40Hz) are attributed to the effect of parasympathetic nervous system, while, the low frequency bands (0.04-0.15 Hz) are attributed to the effect of both sympathetic and parasympathetic nervous systems.

In this study, all patients with spontaneous intracranial bleedings undergo standard treatment and monitoring. This include electrocardiography, arterial blood pressure, and cerebral blood flow using transcranial Doppler sonography. For those who also have intracranial pressure monitoring, the intracranial pressure are also recorded. All these biological signals are exported for wave form analysis. We use frequency analysis, time-frequency analysis, and multiscale entropy to analyze these data. The results of analyses were also correlated to plasma catecholamine levels, proinflammatory markers, as well as the clinical variables. Our aim is to identify predictors of complications and grave outcomes from these biological signals. We also apply the results for future pathophysiological studies.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracranial hemorrhage with radiographical confirmation

Exclusion Criteria:

* Traumatic or undefined mechanisms for intracranial hemorrhage
* Pre-existing cardiac arrythmia
* Patients who had previous histories of intracranial, cardiac, hepatic, renal, or lung diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spontaneous intracranial hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Activity of autonomic nervous activities determined by low frequency and high frequency energies in heart rate variability | 14 days within initial ictus

SECONDARY OUTCOMES:
Presence of vasospasm or not | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Kwang Tu, M.D.., Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Department of Surgery, National Taiwan University Hospital, Taipei
  - Devision of Neurosurgery, National Taiwan University Hospital, Taipei